CLINICAL TRIAL: NCT04560023
Title: Effectiveness of Multimedia Content Exposure in Improving the Experience and Reported Patient Outcomes in Patients Suffering From Acute Mycardial Infarction During the Transfer to Hospital: a Clinical Trial.
Brief Title: Effectiveness of Multimedia Exposure in Patients Transferred to Hospital Suffering From Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cadiz (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Principal Investigator, Sergio Cazorla Calderon, Co-Investigator; PhDc, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ITI-PI-0019-N-17
Record Dates: First submitted 2019-10-20; First posted 2020-09-23 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Myocardial Infarction, Acute; Anxiety State; Emergencies
Keywords: ambulances; video
MeSH Terms: conditions — Myocardial Infarction; Anxiety Disorders; Emergencies

STUDY DESIGN:
Intervention Model Description: Randomisation in blocks will be considered. Software will contain and allocation sequence, in each block, 50% of patients will be allocated in control group (standard practice) and the other 50% will be allocated in the experimental group (multimedia exposure).
Who Masked: Outcomes Assessor
Masking Description: Randomization variable encoding will be blinded for researchers, only known by an external collaborator designed by the main researcher.
  Statistical analysis will be performed by researchers who will be blinded for the assignation to experimental and control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposition to multimedia content (Experimental): Ad hoc design multimedia content in a tablet (video with sound and subtitles).
  Interventions: Other: Exposition to multimedia content
- Standard procedures (No Intervention): Standard procedures.

INTERVENTIONS:
Other: Exposition to multimedia content — Video and images watched on a tablet. Patient could decide which information want to watch.
  Arms: Exposition to multimedia content

SUMMARY:
Randomised clinical trial, single-center, blinded assessment, controlled with standard practice with two-group parallel design.

Eligible patients are those assisted and transferred suffering from ST-Elevation myocardial infarction in an Advanced Life Support ambulance from an public Emergency Medical Service in the Cadiz area (Spain).

Experimental group will watch an ad hoc design multimedia content in a tablet (video with sound and subtitles) during the transfer and control group will be assisted as standard procedures.

Main outcome variables will be conformed by patient reported outcomes (anxiety State, pain and comfort) and patient experience (transfer experience).

DETAILED DESCRIPTION:
Due to intrinsic characteristics of ambulance transport raises stress or anxiety in patients. Moreover, other outcomes such as pain and some specific vital signs are affected. In the last years, empowerment patient strategies have been launched in several clinical settings but none in the ER field.

Main objective Comparative assessment of the effectiveness of multimedia exposure vs standard clinical procedures to improve the experience and patient reported outcomes in patients suffering from ST-Elevation myocardial infarction transferred to hospital in an Advanced Life Support ambulance for a percutaneous coronary intervention (PCI).

Methods Randomised clinical trial, single-center, blinded assessment, controlled with usual practice with two-group parallel design.

Eligible patients are those assisted and transferred suffering from STEMI in an Advance Life Support (ALS) ambulance from public Emergency Medical System in the Cadiz region.

Experimental group will watch multimedia content on a tablet (movie or image with sound) ad hoc designed, control group will be assisted as usual procedures.

Main outcomes will be conformed by informed patient results (anxiety State, pain and comfort) and patient experience (transfer experience).

ELIGIBILITY:
Inclusion Criteria:

* All genders patients.
* Assisted by ALS ambulance.
* Diagnosed with STEMI, "Killip I".
* Transferred by an ambulance to the hospital to receive a percutaneous coronary intervention.
* Informed consent must be signed.
* Conscious and oriented patients.

Exclusion Criteria:

* Sedation and/or assisted ventilation.
* Blinded or visual defects.
* Deafness.
* Severe mental disorders or behavior disorders.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety state | Minute 0.
  Tool State-Trait Anxiety Scale (STAI-E6). Less punctuation means better outcomes. Range 0-18.
Anxiety state change | Minute 10.
  Tool State-Trait Anxiety Scale (STAI-E6). Less punctuation means better outcomes. Range 0-18.
Experience measure of the ambulance service | 1 measure: one week after the patient has been discharge from hospital. Qualitative interview tool.
  Tool Ambulance Patient Reported Experience Measure (APREMS)
Comfort | Minute 0.
  "Kolcaba General Comfort Questionnaire scale". More punctuation means better outcomes. Range 0-10.
Comfort change | Minute 10.
  "Kolcaba General Comfort Questionnaire scale". More punctuation means better outcomes. Range 0-10.

SECONDARY OUTCOMES:
Pain assessment | Minute 0.
  Analogic Pain Scale. Less punctuation means better outcomes. Range 0-10.
Pain assessment change | Minute 10.
  Analogic Pain Scale. Less punctuation means better outcomes. Range 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Paloma, PhD, Principal Investigator — Universidad Cádiz
Locations (1):
- Universidad de Cádiz, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No